CLINICAL TRIAL: NCT01195545
Title: Veritas Laparoscopic PEH Repair Pilot Trial
Brief Title: Veritas Laparoscopic Paraesophageal Hiatal Hernia (PEH) Repair Pilot Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Synovis Surgical Innovations (Industry)
Responsible Party: Principal Investigator, Brant Oelschlager, Professor and Chief of General Surgery, Surgery, General Surgery Division, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38048
Record Dates: First submitted 2010-09-02; First posted 2010-09-06 (Estimated); Results first posted 2018-07-10 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-06

CONDITIONS: Hiatal Hernia
Keywords: Veritas® Collagen Matrix, Hiatal hernia
MeSH Terms: conditions — Hernia, Hiatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Veritas Mesh in Hernia Repair (Experimental): Subjects undergoing laparoscopic paraesophageal hiatal hernia repair using a bovine pericardium mesh (BP) (Veritas® Collagen Matrix, Synovis ®, St. Paul MN) as a reinforcing material during repair.
  Interventions: Device: Veritas® Collagen Matrix

INTERVENTIONS:
Device: Veritas® Collagen Matrix — biological mesh in hernia repair

SUMMARY:
This is an investigator initiated pilot study to observe the short-term outcomes (a follow-up period of up to six months) of patients who undergo a laparoscopic paraesophageal Hiatal hernia (PEH) repair using the Veritas® Collagen Matrix brand biological mesh. This is a preliminary study at the University of Washington.

A PEH occurs when the stomach protrudes through the diaphragm next to the esophagus. The chance of recurrence of a Hiatal hernia after laparoscopic PEH repair is between 20-40% within 6 months.During laparoscopic PEH repair, a mesh-type product is used as a scaffold. The mesh serves as a reinforcing material during the surgical repair. It is cut to the appropriate size needed for the hernia and sutured to the surrounding diaphragmatic tissue. There are many different types of meshes available on the market, and vary in the degree of manageability, strength, and adherence.

Although surgical meshes work on the same principal, the variance between materials may affect patient outcomes. There is evidence that a biologic mesh, specifically one derived from Small Intestinal Submucosa (SIS), decreases the short-term (6-month) recurrence rates compared to a synthetic mesh or another type of biologic mesh. A biologic mesh, serving as a scaffold, will be replaced by the patient's own tissue after about 6 months. Theoretically, this would prevent the possible complications associated with synthetic mesh including mesh erosion into the esophagus or stricture of the esophagus.

There are some case series showing similar short-term results between the different biologic meshes, but there is no direct comparative data.

ELIGIBILITY:
Inclusion Criteria:

A. Subjects must have a documented symptomatic paraesophageal hernia that:

* 1. Is greater than 5 cm hiatal hernia on Upper Gastrointestinal (UGI) series
* 2. Has evidence that the stomach or other viscera is present in the hernia and does not spontaneously reduce from the mediastinum
* 3. Has significant symptoms or signs of a paraesophageal hernia: heartburn, dysphagia, chest pain, shortness of breath, post-prandial abdominal pain, early satiety, odynophagia or chronic anemia

B. Consenting adult ≥18 years ~ documentation of informed consent will be recorded in the research records

C. Must be able to participate in follow-up evaluations (subjects must be fully cognitive)

D. Has a telephone

E. Free of cognitive or speech impairment

Exclusion Criteria:

A. Previous operation of the esophagus or stomach

B. Associated gastrointestinal diseases that require extensive medical or surgical intervention that might interfere with quality of life assessment (e.g. Crohn's disease)

C. Emergent operation for acute volvulus (twisting/rotation of the bowel leading to obstruction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brant K. Oelschlager, M.D., Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Veritas Mesh in Hernia Repair: Subjects undergoing laparoscopic paraesophageal hiatal hernia repair using a bovine pericardium mesh (BP) (Veritas® collagen matrix, Synovis®, St. Paul MN) as a reinforcing material during the repair.
Period: Overall Study
Arm/Group | Veritas Mesh in Hernia Repair
Started | 20
Completed | 16
Not Completed | 4
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Population: Subjects undergoing laparoscopic paraesophageal hiatal hernia repair using a bovine pericardium mesh (BP) (Veritas® collagen matrix, Synovis®, St. Paul MN) as a reinforcing material during the repair.
Arm/Group | Veritas Mesh in Hernia Repair
Number analyzed (Participants) | 20
Age, Customized [Median (Full Range); unit: years]
  Age | 66 [47 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 20
BMI [Median (Full Range); unit: kg/m^2] | 28.7 [21.9 to 40.2]

OUTCOME MEASURES:

1. Primary Outcome: Recurrence Rate of Hiatal Hernia Rate Based on Upper Gastrointestinal (UGI) Series
Description: Number of subjects experiencing recurrence greater than 2cm as well as 5cm post surgery.
Time Frame: 6 months post procedure
Population: 6 months post-op follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Veritas Mesh in Hernia Repair
Number analyzed (Participants) | 16
Participants
  Recurrence >2cm | 6
  Recurrence >5cm | 2
  No evidence of recurrence. | 8

2. Secondary Outcome: Pre and Post-operative Symptoms
Description: Heartburn frequency Pre and Post-operative was measured using the Paraesophagel Hernia Patient Questionnaire-Visual analog score (VAS). The VAS measures subjective characteristics that specify the respondents level of agreement to a statement. In this questionnaire, the patient indicated how frequent they had Heartburn. The Heartburn frequency measurement scale: 0=Never, 1=once/month,2=once/week,3=once/day,4=several/day. The lower the VAS score the better the outcome meaning less episodes of Heartburn.
  The Heartburn VAS score was measured pre-operative and post-operative. The comparison of Heartburn VAS score pre-operative and post-operative indicated that participants experienced Improvement and No Improvement.
Time Frame: Pre-surgery and 6 month follow up
Population: Pre-surgery and at a median follow up 6 months month (range 3 - 10 months)
Measure: Count of Participants; unit: Participants
Arm/Group | Veritas Mesh in Hernia Repair
Number analyzed (Participants) | 16
Participants
  With Improvement of Heartburn | 15
  No Improvement of Heartburn | 1

3. Secondary Outcome: Pre and Post-operative Symptoms
Description: Regurgitation frequency Pre and Post-operative was measured using the Paraesophagel Hernia Patient Questionnaire-Visual analog score (VAS). The VAS measures subjective characteristics that specify the respondents level of agreement to a statement. In this questionnaire, the patient indicated how frequent they had Regurgitation. The Regurgitation frequency measurement scale: 0=Never, 1=once/month,2=once/week,3=once/day,4=several/day. The lower the VAS score the better the outcome meaning less episodes of Regurgitation.
  The Regurgitation VAS score was measured pre-operative and post-operative. The comparison of Regurgitation VAS score pre-operative and post-operative indicated that participants experienced Improvement and No Improvement.
Time Frame: Pre-surgery and 6 month follow up
Population: Pre-surgery an at median follow up of 6 month (3-6 month)
Measure: Count of Participants; unit: Participants
Arm/Group | Veritas Mesh in Hernia Repair
Number analyzed (Participants) | 16
Participants
  Improvement in regurgitation | 11
  No improvement in regurgitation | 5

4. Secondary Outcome: Pre and Post-operative Symptoms
Description: Dysphagia frequency Pre and Post-operative was measured using the Paraesophagel Hernia Patient Questionnaire-Visual analog score (VAS). The VAS measures subjective characteristics that specify the respondents level of agreement to a statement. In this questionnaire, the patient indicated how frequent they had Dysphagia. The Dysphagia frequency measurement scale: 0=Never, 1=once/month,2=once/week,3=once/day,4=several/day. The lower the VAS score the better the outcome meaning less episodes of Dysphagia.
  The Dysphagia VAS score was measured pre-operative and post-operative. The comparison of Dysphagia VAS score pre-operative and post-operative indicated that some participants experienced Improvement and others worsen.
Time Frame: Pre-surgery and 6 month follow up
Population: Pre-surgery and a median of 6 month follow up (3-6months)
Measure: Count of Participants; unit: Participants
Arm/Group | Veritas Mesh in Hernia Repair
Number analyzed (Participants) | 16
Participants
  Dysphagia Improved | 14
  Dysphagia worsen | 2

ADVERSE EVENTS:
Groups:
- Experimental: Subjects undergoing laparoscopic paraesophageal hiatal hernia repair using a bovine pericardium mesh (BP) (Veritas® collagen matrix, Synovis®, St. Paul MN) as a reinforcing material during the repair.
Arm/Group | Experimental
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes